CLINICAL TRIAL: NCT01433458
Title: A Single-dose, Open-label Parallel Study to Assess the Pharmacokinetics of RLX030 in Subjects With Mild, Moderate and Severe Hepatic Impairment Compared to Healthy Control Subjects
Brief Title: Pharmacokinetics of RLX030 in Subjects With Mild, Moderate and Severe Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRLX030A2101; 2011-001596-39 (EudraCT Number)
Record Dates: First submitted 2011-08-09; First posted 2011-09-14 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2013-01

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; healthy volunteers; RLX030; pharmacokinetics

ARMS (4):
- RLX030: Group 1 mild hepatic impairment (Experimental): Patients with mild hepatic impairment will receive a single IV 24 hour infusion of RLX030
  Interventions: Drug: RLX030A
- RLX030: Group 2 moderate hepatic impairment (Experimental): Patients with moderate hepatic impairment will receive a single IV 24 hour infusion of RLX030
  Interventions: Drug: RLX030A
- RLX030: Group 3 severe hepatic impairment (Experimental): Patients with severe hepatic impairment will receive a single IV 24 hour infusion of RLX030
  Interventions: Drug: RLX030A
- RLX030: Group 4 - healthy volunteers (Active Comparator): Participants will receive a single IV 24 hour infusion of RLX030. This group will consist of 3 sub-groups to match patients of groups 1, 2and 3.
  Interventions: Drug: RLX030A

INTERVENTIONS:
Drug: RLX030A — RLX030 is administered as a continuous 24 hour infusion

SUMMARY:
This study will assess the pharmacokinetics of RLX030 during and after administration in subjects with mild to severe hepatic impairment and matched healthy control subjects.

20 to 24 patients and 20 to 24 healthy subjects will be enrolled.

ELIGIBILITY:
Inclusion criteria:

* All subjects:

  • Female subjects must be of non-child bearing potential OR use an effective method of contraception and sexually active males must use a condom during intercourse while taking the drug and for 5 half-lives after stopping treatment
* Subjects with hepatic impairment:

  * Subjects must have either mild, moderate or severe hepatic impairment

Exclusion criteria:

* All subjects

  * Hepatic impairment due to non-liver disease
  * Use of other investigational drugs at time of enrollment
  * History of malignancy of any organ system
  * Donation or loss of 400 mL or more of blood or plasma within 8 weeks prior to initial dosing
  * Hemoglobin levels below 10.0 g/dL at screening or baseline
* Subjects with hepatic impairment:

  * Presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the patient at undue risk
  * Treatment with any cytostatic drug, vasodilator, autonomic alpha blocker or B2 agonist
  * Any surgical or medical condition other than hepatic impairment which might significantly alter the distribution or excretion of drugs

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to infinity (AUCinf) | Up to Day 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Up to Day 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030
Serum concentration at 24 hour (C24h) after administration | Upto Day 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030

SECONDARY OUTCOMES:
Number of patients with adverse events, serious adverse events and death | Day 15
  Monitoring of adverse events, serious adverse events and death from screening to end of study
Determination of the presence and quantification of anti-RLX030 antibodies | Day 1 (prior to administration) and Day 15 end of study
  Blood will be collected and serum analyzed for the presence of antiRLX030 antibodies. Anti-RLX030 antibodies will be evaluated in serum in a validated four-tiered assay approach
Mean residence time [MRT] of RLX030 | screening, days 1, 2, 3, 4 and 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030
Terminal elimination half life (T ½) of RLX030 | screening, days 1, 2, 3, 4 and 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030
Systemic clearance of RLX030 from serum (CL) | screening, days 1, 2, 3, 4 and 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030
Volume of distribution at steady state (Vss) | screening, days 1, 2, 3, 4 and 15
  Blood samples will be collected during screening, days 1 through 4 and then on Day 15 for the determination of serum concentrations of RLX030

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Grünstadt, Germany
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- [Derived] Kobalava Z, Villevalde S, Kotovskaya Y, Hinrichsen H, Petersen-Sylla M, Zaehringer A, Pang Y, Rajman I, Canadi J, Dahlke M, Lloyd P, Halabi A. Pharmacokinetics of serelaxin in patients with hepatic impairment: a single-dose, open-label, parallel group study. Br J Clin Pharmacol. 2015 Jun;79(6):937-45. doi: 10.1111/bcp.12572. PMID 25511105
- See also: Results for CRLX030A2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7565